CLINICAL TRIAL: NCT03280849
Title: Chitosan Scaffold for Sellar Floor Repair in Endoscopic Endonasal Transsphenoidal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Ivan Segura Duran, M.D., University of Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI.064.2015
Record Dates: First submitted 2017-09-04; First posted 2017-09-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Csf Leakage
Keywords: chitosan; endoscopic; sellar tumor; biomaterials; transphenoidal
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Intervention Model Description: Use of a novel bilaminar chitosan scaffold in the repair of the sellar floor after an endoscopic endonasal transsphenoidal surgery for a suspected hipofisary macroadenoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with bilaminar chitosan implant (Experimental): A 65 year old woman, right handed, started with progressive bilateral visual loss in her temporal field, over 10 months, she underwent an MRI and it was found a sellar lesion that compressed the optic chiasm, an endoscopic endonasal transsphenoidal surgery was done for the resection of the lesion, using a novel bilaminar chitosan scaffold to assist the closure of the sellar floor.
  Interventions: Other: Implant of bilaminar chitosan scaffold

INTERVENTIONS:
Other: Implant of bilaminar chitosan scaffold — The patient underwent endoscopic endonasal transsphenoidal surgery for resection of the sellar lesion, under the direct visualization, the lesion appeared redish and soft with moderately bleeding, a sample was taken for pathology and the remaining is extracted without complications, then the scaffold is implanted in the site of the bone defect in the sphenoid sinus, due to its moldable nature, it was easily set, covering the entire extension of the defect, a fat graft was set in the sphenoid sinus covering the bilaminar chitosan membrane, then fibrin sealant was used for hemostatic control and a nasal packing was set in both nostrils for finalize the procedure.
  Other Names: Endoscopic endonasal transphenoidal surgery

SUMMARY:
A 65 year old female participant , right handed, started with progressive bilateral visual loss in her temporal field, over 10 months, the participant underwent an MRI and it was found a sellar lesion that compressed the optic chiasm, an endoscopic endonasal transsphenoidal surgery was done for the resection of the lesion, using a novel bilaminar chitosan scaffold to assist the closure of the sellar floor. After a follow up of 2 years the participant returned to its normal visual function, without evidence of the sellar lesion on the postoperative MRI, and without complications.

DETAILED DESCRIPTION:
Introduction This case describe the use of a novel bilaminar chitosan scaffold in the repair of the sellar floor after an endoscopic endonasal transsphenoidal surgery for a suspected hipofisary macroadenoma, the use of chitosan as a scaffold has been described in several preclinical studies and tested in tissue bioengineering of bone, neural tissue and soft tissue, in the case of bone tissue, several studies demonstrated its potential due to its biocompatibility, osteinductive and osteoconductive features, but there is a lack of clinical trials demonstrating this characteristics in the clinical setting. One of the most common complications for the neurosurgeons after an endoscopic endonasal transsphenoidal surgery is the CSF leak, depending on the technique and the reconstruction used for the sellar floor this complication could be presented from 5% to 75%of the cases, leading to complications such infections and pneumoencephalus, representing a great risk for comorbidities, longer recovery times and hospital costs, due to this challenges in the repair of the sellar floor,the investigators intent to approach the problematic with a chitosan scaffold for its characteristics in bone regeneration. The setting of a bioactive membrane in the defect of the surgery could be useful for a stronger and more suitable closure of the sellar floor.

Case description A 65 years old female participant, right handed, came to the neurosurgery consultation with progressive bilateral visual loss in her temporal fields, with predominance in the left eye over 10 months, two weeks before her admission the participant reported a sudden loss of consciousness, prompting her to go to the hospital. In her clinical examination, the participant was alert and oriented x3, normal cranial nerves examination except for decrease visual acuity by 20/200 in her left eye, 20/80 in her right eye, bitemporal hemianopia and mild primary athropy of the optic disc in the left eye, the gait and the motor and sensitive examination was normal. The laboratory studies showed a LH: 0.22 and prolactine: 53.7 .In the contrasted preoperative brain MRI, it was found a sellar lesion, hypointense in T1 but hyperintense in T2 signal with enhancing of the periphery after the infusion of gadolinium, the lesion presented extension to the sphenoid sinus, paraselar space without involvement of the carotids and supraselar with displacement of the optic chiasm. The participant underwent endoscopic endonasal transsphenoidal surgery for resection of the sellar lesion, under the direct visualization, the lesion appeared redish and soft with moderately bleeding, a sample was taken for pathology and the remaining is extracted without complications, then the scaffold is implanted in the site of the bone defect in the sphenoid sinus, due to its moldable nature, it was easily set, covering the entire extension of the defect, a fat graft was set in the sphenoid sinus covering the bilaminar chitosan membrane, then fibrin sealant was used for hemostatic control and a nasal packing was set in both nostrils for finalize the procedure. In the postoperative there was not complication and after a few days the participant was discharged with notable clinical improvement, after one month of follow up the participant recovered her visual acuity and the participant did not refer any symptom, the participant underwent a post operative brain MRI, where it is observed a gross total resection and good closure of the sellar floor, without signs of rejection or inflammation in the zone with the chitosan scaffold.

Materials and methods for the bilaminar chitosan scaffold The bilaminar implant is constitute by two types of different structures, one of the membranes presents a flat-smooth structure, the other membrane has a tridimensional-porous structure, each of the physical-chemical characteristics given to the membranes, was in function of the biological effect pretended in the effector tissue.

The two types of membranes, synthetized for the elaboration of the bilaminar implant, were elaborated with biomedical grade chitosan of medium molecular weight with 75-85% of deacetylation in powder presentation from the brand Sigma Aldrich®, U.S.A.

In the case of the membrane with flat-smooth structure, it was synthetized from a chitosan solution at 2%, the dissolution medium was diluted acetic acid (Sigma Aldrich®, U.S.A); In order to acquired a suitable solubilisation, the mix was set on a magnetic stirrer for 1 hour, posteriorly the solution was brought under the action of a sonicator at 28oc for 2 hours, until the air bubbles formed by the stirrer were completely eliminated.

For the membrane with the tridimensional-porous structure, it was synthetized from a chitosan solution at 4%, the dissolution medium was diluted acetic acid (Sigma Aldrich®, U.S.A); for a suitable solubilisation, the mix was set on a magnetic stirrer for 4 hours, afterward the solution was brought under the action of a sonicator at 28oc for 2 hours, until the air bubbles formed by the stirrer were completely eliminated.

Once the solutions were elaborated, for the synthesis of the two membranes (the flat-smooth and the tridimensional-porous) both were set in a constant quantity of ml/cm2 in a Petri dish, in the case of the flat-smooth membrane, it was brought under a procedure of drying with 98% of humidity loss and for the tridimensional-porous, a procedure of phase separating was termical induced.

When both membranes are already elaborated, it is proceed to synthetize the bilaminar implant, the membranes are combined using a solution of chitosan acetate at 2%, that was distributed uniformly between both membranes to create a sandwich structure, consecutively the ensemble was put in a Petri dish and the cover was set inverted in the superior aspect of petri dish. It was set for drying for 24 hours at room temperature and then it was precipitated in a solution of sodium hydroxide 1N, following the same indications used for each membrane separately.

ELIGIBILITY:
Inclusion Criteria:

* male/female patient candidate for an endoscopic endonasal transphenoidal surgery, who need repair of the sellar floor as part of the surgical procedure.

Exclusion Criteria:

* Diabetes, heart diseases, immunological diseases, infectious diseases, bone diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Brain MRI with and without contrast | 1 day preoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the preoperative tumor size
Brain MRI with and without contrast | 1 day postoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the postoperative tumor size
Head CT scan | 1 month postoperative
  Bone window was used to see the repair of bone defect after surgery
Brain MRI with and without contrast | 1 month postoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the postoperative tumor
Brain MRI with and without contrast | 6 months postoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the postoperative tumor
Brain MRI with and without contrast | 1 year postoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the postoperative tumor
Brain MRI with and without contrast | 2 years postoperative
  Axial-coronal-sagittal MRI in T1,T2 signals-measure of the postoperative tumor
Head CT scan | 6months postoperative
  Bone window was used to see the repair of bone defect after surgery
Head CT scan | 1 year postoperative
  Bone window was used to see the repair of bone defect after surgery
Head CT scan | 2 years postoperative
  Bone window was used to see the repair of bone defect after surgery

SECONDARY OUTCOMES:
Visual field test | 1 day preoperative, follow up: 1 day postoperative, 15 days postoperative, 1 month postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
  visual field testing looking for compression of optic chiasm
Snellen test | 1 day preoperative, follow up: 1 day postoperative, 15 days postoperative, 1 month postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
  visual acuity testing
Glasgow scale | 1 day preoperative, follow up :1 day postoperative, 15 days postoperative, 1 month postoperative, 6 months postoperative, 1 year postoperative, 2 years postoperative.
  level of consciousness
Endocrinological panel | 1 day preoperative, follow up : 1 day postoperative, 15 days postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  evaluation of hipofisary function
Blood cell count | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  For evaluation of any inflammatory reaction or infection before or after the procedure
acute phase reactans | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  For evaluation of any inflammatory reaction or infection before or after the procedure
blood electrolytesand | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  evaluation of renal function and as requirement for surgery
liver function test | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  evaluation of liver function and as requirement for surgery
coagulation test | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  secondary evaluation of liver function, inflammatory reaction or infection before and after the procedure and as requirement for surgery.
seric creatinine | 1 day preoperative, follow up: 1 day postoperative , 1 month postoperative, 6 months postoperative,1 year postoperative, 2 years postoperative
  evaluation of renal function and as requirement for surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ramos Zuñiga, M.D. PhD, Study Chair — University of Guadalajara; Brenda Vega Ruiz, PhD, Principal Investigator — University of Guadalajara; Ivan Segura Duran, M.D., Principal Investigator — University of Guadalajara
Locations (1):
- Departamento de neurociencias, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
complete MRI sequences, laboratory studies, visual field tests, complete biomaterial patent registration , clinical reports.

REFERENCES:
- [Background] Gobin AS, Butler CE, Mathur AB. Repair and regeneration of the abdominal wall musculofascial defect using silk fibroin-chitosan blend. Tissue Eng. 2006 Dec;12(12):3383-94. doi: 10.1089/ten.2006.12.3383. PMID 17518675
- [Background] Paulo NM, de Brito e Silva MS, Moraes AM, Rodrigues AP, de Menezes LB, Miguel MP, de Lima FG, de Morais Faria A, Lima LM. Use of chitosan membrane associated with polypropylene mesh to prevent peritoneal adhesion in rats. J Biomed Mater Res B Appl Biomater. 2009 Oct;91(1):221-7. doi: 10.1002/jbm.b.31393. PMID 19399842
- [Background] Udpa N, Iyer SR, Rajoria R, Breyer KE, Valentine H, Singh B, McDonough SP, Brown BN, Bonassar LJ, Gao Y. Effects of chitosan coatings on polypropylene mesh for implantation in a rat abdominal wall model. Tissue Eng Part A. 2013 Dec;19(23-24):2713-23. doi: 10.1089/ten.TEA.2012.0739. Epub 2013 Aug 21. PMID 23859182
- [Background] Tchemtchoua VT, Atanasova G, Aqil A, Filee P, Garbacki N, Vanhooteghem O, Deroanne C, Noel A, Jerome C, Nusgens B, Poumay Y, Colige A. Development of a chitosan nanofibrillar scaffold for skin repair and regeneration. Biomacromolecules. 2011 Sep 12;12(9):3194-204. doi: 10.1021/bm200680q. Epub 2011 Aug 1. PMID 21761871
- [Background] Stippler M, Gardner PA, Snyderman CH, Carrau RL, Prevedello DM, Kassam AB. Endoscopic endonasal approach for clival chordomas. Neurosurgery. 2009 Feb;64(2):268-77; discussion 277-8. doi: 10.1227/01.NEU.0000338071.01241.E2. PMID 19190456
- [Background] Gardner PA, Kassam AB, Snyderman CH, Carrau RL, Mintz AH, Grahovac S, Stefko S. Outcomes following endoscopic, expanded endonasal resection of suprasellar craniopharyngiomas: a case series. J Neurosurg. 2008 Jul;109(1):6-16. doi: 10.3171/JNS/2008/109/7/0006. PMID 18590427
- [Background] Greenfield JP, Anand VK, Kacker A, Seibert MJ, Singh A, Brown SM, Schwartz TH. Endoscopic endonasal transethmoidal transcribriform transfovea ethmoidalis approach to the anterior cranial fossa and skull base. Neurosurgery. 2010 May;66(5):883-92; discussion 892. doi: 10.1227/01.neu.0000368395.82329.c4. PMID 20414977
- [Background] Gardner PA, Kassam AB, Thomas A, Snyderman CH, Carrau RL, Mintz AH, Prevedello DM. Endoscopic endonasal resection of anterior cranial base meningiomas. Neurosurgery. 2008 Jul;63(1):36-52; discussion 52-4. doi: 10.1227/01.NEU.0000335069.30319.1E. PMID 18728567
- [Result] Simoes MJ, Gartner A, Shirosaki Y, Gil da Costa RM, Cortez PP, Gartner F, Santos JD, Lopes MA, Geuna S, Varejao AS, Mauricio AC. In vitro and in vivo chitosan membranes testing for peripheral nerve reconstruction. Acta Med Port. 2011 Jan-Feb;24(1):43-52. Epub 2011 Feb 28. PMID 21672441
- [Result] Meyer C, Stenberg L, Gonzalez-Perez F, Wrobel S, Ronchi G, Udina E, Suganuma S, Geuna S, Navarro X, Dahlin LB, Grothe C, Haastert-Talini K. Chitosan-film enhanced chitosan nerve guides for long-distance regeneration of peripheral nerves. Biomaterials. 2016 Jan;76:33-51. doi: 10.1016/j.biomaterials.2015.10.040. Epub 2015 Oct 21. PMID 26517563
- [Result] Zhao Y, Wang Y, Gong J, Yang L, Niu C, Ni X, Wang Y, Peng S, Gu X, Sun C, Yang Y. Chitosan degradation products facilitate peripheral nerve regeneration by improving macrophage-constructed microenvironments. Biomaterials. 2017 Jul;134:64-77. doi: 10.1016/j.biomaterials.2017.02.026. Epub 2017 Feb 22. PMID 28456077
- [Result] Ghasemi Hamidabadi H, Rezvani Z, Nazm Bojnordi M, Shirinzadeh H, Seifalian AM, Joghataei MT, Razaghpour M, Alibakhshi A, Yazdanpanah A, Salimi M, Mozafari M, Urbanska AM, Reis RL, Kundu SC, Gholipourmalekabadi M. Chitosan-Intercalated Montmorillonite/Poly(vinyl alcohol) Nanofibers as a Platform to Guide Neuronlike Differentiation of Human Dental Pulp Stem Cells. ACS Appl Mater Interfaces. 2017 Apr 5;9(13):11392-11404. doi: 10.1021/acsami.6b14283. Epub 2017 Mar 27. PMID 28117963
- [Result] Rodriguez-Vazquez M, Vega-Ruiz B, Ramos-Zuniga R, Saldana-Koppel DA, Quinones-Olvera LF. Chitosan and Its Potential Use as a Scaffold for Tissue Engineering in Regenerative Medicine. Biomed Res Int. 2015;2015:821279. doi: 10.1155/2015/821279. Epub 2015 Oct 4. PMID 26504833
- [Result] Sandoval-Sanchez JH, Ramos-Zuniga R, de Anda SL, Lopez-Dellamary F, Gonzalez-Castaneda R, Ramirez-Jaimes Jde L, Jorge-Espinoza G. A new bilayer chitosan scaffolding as a dural substitute: experimental evaluation. World Neurosurg. 2012 Mar-Apr;77(3-4):577-82. doi: 10.1016/j.wneu.2011.07.007. Epub 2011 Nov 7. PMID 22120335
- [Result] Nawrotek K, Marqueste T, Modrzejewska Z, Zarzycki R, Rusak A, Decherchi P. Thermogelling chitosan lactate hydrogel improves functional recovery after a C2 spinal cord hemisection in rat. J Biomed Mater Res A. 2017 Jul;105(7):2004-2019. doi: 10.1002/jbm.a.36067. Epub 2017 Apr 12. PMID 28324618
- [Result] Mota J, Yu N, Caridade SG, Luz GM, Gomes ME, Reis RL, Jansen JA, Walboomers XF, Mano JF. Chitosan/bioactive glass nanoparticle composite membranes for periodontal regeneration. Acta Biomater. 2012 Nov;8(11):4173-80. doi: 10.1016/j.actbio.2012.06.040. Epub 2012 Jul 5. PMID 22771458
- [Result] Azevedo AS, Sa MJ, Fook MV, Neto PI, Sousa OB, Azevedo SS, Teixeira MW, Costa FS, Araujo AL. Use of chitosan and beta-tricalcium phosphate, alone and in combination, for bone healing in rabbits. J Mater Sci Mater Med. 2014 Feb;25(2):481-6. doi: 10.1007/s10856-013-5091-2. Epub 2013 Nov 17. PMID 24243224
- [Result] Fan J, Park H, Lee MK, Bezouglaia O, Fartash A, Kim J, Aghaloo T, Lee M. Adipose-derived stem cells and BMP-2 delivery in chitosan-based 3D constructs to enhance bone regeneration in a rat mandibular defect model. Tissue Eng Part A. 2014 Aug;20(15-16):2169-79. doi: 10.1089/ten.TEA.2013.0523. Epub 2014 May 9. PMID 24524819
- [Result] Zhao F, Yin Y, Lu WW, Leong JC, Zhang W, Zhang J, Zhang M, Yao K. Preparation and histological evaluation of biomimetic three-dimensional hydroxyapatite/chitosan-gelatin network composite scaffolds. Biomaterials. 2002 Aug;23(15):3227-34. doi: 10.1016/s0142-9612(02)00077-7. PMID 12102194
- [Result] Liuyun J, Yubao L, Chengdong X. A novel composite membrane of chitosan-carboxymethyl cellulose polyelectrolyte complex membrane filled with nano-hydroxyapatite I. Preparation and properties. J Mater Sci Mater Med. 2009 Aug;20(8):1645-52. doi: 10.1007/s10856-009-3720-6. Epub 2009 Mar 20. PMID 19301105
- [Result] Zhang J, Wang C, Wang J, Qu Y, Liu G. In vivo drug release and antibacterial properties of vancomycin loaded hydroxyapatite/chitosan composite. Drug Deliv. 2012 Jun-Jul;19(5):264-9. doi: 10.3109/10717544.2012.704093. PMID 22823893
- [Result] Pu XM, Yao QQ, Yang Y, Sun ZZ, Zhang QQ. In vitro degradation of three-dimensional chitosan/apatite composite rods prepared via in situ precipitation. Int J Biol Macromol. 2012 Dec;51(5):868-73. doi: 10.1016/j.ijbiomac.2012.07.008. Epub 2012 Jul 16. PMID 22800729
- [Result] Kim SB, Kim YJ, Yoon TL, Park SA, Cho IH, Kim EJ, Kim IA, Shin JW. The characteristics of a hydroxyapatite-chitosan-PMMA bone cement. Biomaterials. 2004 Nov;25(26):5715-23. doi: 10.1016/j.biomaterials.2004.01.022. PMID 15147817
- [Result] Teng SH, Lee EJ, Wang P, Shin DS, Kim HE. Three-layered membranes of collagen/hydroxyapatite and chitosan for guided bone regeneration. J Biomed Mater Res B Appl Biomater. 2008 Oct;87(1):132-8. doi: 10.1002/jbm.b.31082. PMID 18395825
- See also: website of our institute of traslational neurosciences — http://www.cucs.udg.mx/instituto-de-neurociencias-traslacionales
- See also: website of our center — http://www.cucs.udg.mx/general/departamento-de-neurociencias
- See also: website of our hospital facilities — http://www.hcg.udg.mx